CLINICAL TRIAL: NCT06265376
Title: A Single-site Randomized Controlled Trial of an Patient Educational Video to Improve Postoperative Pain and Overall Recovery Satisfaction After Laparoscopic Hysterectomy Benign Indication
Brief Title: Do Patient Educational Videos Improve Pain and Recovery After Laparoscopic Hysterectomy?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benaroya Research Institute (Other)
Responsible Party: Principal Investigator, Megan Loring, MD, Gynecologist, Benaroya Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB22-046
Record Dates: First submitted 2024-01-04; First posted 2024-02-20 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Video Intervention (Experimental): Participants have been randomly selected into this arm to receive intervention via the educational video in addition to regular treatment and recovery options.
  Interventions: Behavioral: Educational Video
- No Intervention (No Intervention): Participants have been randomly selected into this arm to not receive intervention and continue with regular treatment and recovery options.

INTERVENTIONS:
Behavioral: Educational Video — A recorded educational video will be presented to the patient prior to meeting with the provider at the presurgical meeting
  Arms: Educational Video Intervention

SUMMARY:
The use of multi-model patient education has been used in a variety of medical specialties to educate patients on expectations for various medical procedures and improve patients' understanding of their own health care. However, it is unknown what type of audio and/or visual materials work best in a given clinical setting. By surveying overall pain/post-operative recovery satisfaction we can measure how well our video intervention educates and reinforces post-operative management at home when compared to the current method of education that patients receive at the pre-operative visit prior to laparoscopic hysterectomy at this institution.

ELIGIBILITY:
Inclusion Criteria:

* 18y/o or older
* planned for a laparoscopic hysterectomy for benign indications

Exclusion Criteria:

* inability to consent
* language other than English
* conversion to laparotomy, vNOTES (a type of laparoscopic assisted vaginal hysteroectomy)
* vaginal hysterectomy
* chronic opioid use prior to surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2024-04-28 (Actual); Study Completion 2024-04-28 (Actual)

PRIMARY OUTCOMES:
Overall satisfaction score (5 point Likert scale) with post operative pain control after laparoscopic hysterectomy | Within 10 days post surgery
  To determine if video education on post-operative pain management and expectations can improve patients' overall satisfaction with post operative pain control after laparoscopic hysterectomy

SECONDARY OUTCOMES:
Pain score at the time of survey completion (0=no pain 10=worst pain | Within 10 days post surgery
  To determine if video education on post-operative pain management and expectations improves patient post operative pain scores at the time of post-op phone call
Average pain score for the first 7 days as perceived by the patients (likert scale) | Within 10 days post surgery
  To determine if video education on post-operative pain management and expectations improves patient perceived post operative pain control throughout the first 7 day post-op
Number of post-op phone calls received | Within 10 days post surgery
  To determine if video education on post-operative pain management and expectations decreases the number of post- operative phone calls received by providers during the first week post-op
Number of post-op emergency room visits | Within 10 days post surgery
  To determine if video education on post-operative pain management and expectations decreases the number of post- operative emergency room visits by patients during the first week post-op
Number of readmissions | Within 10 days post surgery
  To determine if video education on post-operative pain management and expectations decreases the number of postoperative readmissions by patients during the first week post-op
Number of patients with steri-strips still in place | Within 10 days post surgery
  To determine if video education on post-operative pain management and expectations decreases the number of patients who have not removed their steri-strips by day 7
Number opioids taken since surgery | Within 10 days post surgery
  To determine if video education on post-operative pain management and expectations decreased the number of narcotics used post-operatively
Overall satisfaction with pre-operative education regarding surgery (5 point Likert scale) | Within 10 days post surgery
  To determine if video education on post-operative pain management and expectations improves overall satisfaction with pre-operative education regarding surgery
ding surgery (5 point likert scale) Overall satisfaction with educations regarding what to expect post-operatively (5 point Likert scale) | Within 10 days post surgery
  To determine if video education on post-operative pain management and expectations improves overall satisfaction with educations regarding what to expect post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Megan Loring, MD, Principal Investigator — Virginia Mason Medical Center
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States